CLINICAL TRIAL: NCT01270464
Title: A 16-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Reslizumab (0.3 or 3.0 mg/kg) as Treatment for Patients (12-75 Years of Age) With Eosinophilic Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety of Reslizumab (0.3 or 3.0 mg/kg) as Treatment for Patients (12-75 Years of Age) With Eosinophilic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C38072/3081; 2010-023342-67 (EudraCT Number)
Record Dates: First submitted 2010-12-29; First posted 2011-01-05 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — reslizumab; Antibodies, Monoclonal, Humanized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered intravenously (iv) once every 4 weeks, for a total of 4 doses.
  Interventions: Drug: Placebo
- Reslizumab - 0.3 mg/kg (Experimental): 0.3 mg/kg, administered intravenously (iv) once every 4 weeks, for a total of 4 doses
  Interventions: Drug: Reslizumab
- Reslizumab - 3.0 mg/kg (Experimental): 3.0 mg/kg, administered intravenously (iv) once every 4 weeks, for a total of 4 doses.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — 3.0 mg/kg or 0.3 mg/kg doses administered intravenously (iv) by qualified site personnel once every 4 weeks, for a total of 4 doses.
  Other Names: Cinquil; humanized monoclonal antibody; CEP-38072
  Arms: Reslizumab - 0.3 mg/kg; Reslizumab - 3.0 mg/kg
Drug: Placebo — Placebo administered by iv infusion by qualified study personnel every 4 weeks for a total of 4 doses.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether reslizumab, at a dosage of 0.3 or 3.0 mg/kg administered once every 4 weeks for a total of 4 doses, is more effective than placebo in improving lung function in patients with eosinophilic asthma as assessed by the overall change from baseline in forced expiratory volume in 1 second (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female, 12 through 75 years of age, with a previous diagnosis of asthma. Patients 12 through 17 years of age are excluded from participating in Argentina.
* The patient has an ACQ score of at least 1.5.
* The patient has airway reversibility of at least 12% to beta-agonist administration at screening.
* The patient is currently taking fluticasone at a dosage of at least 440 μg daily (or equivalent). Patients' baseline asthma therapy regimens (including but not limited to inhaled corticosteroids, leukotriene antagonists, 5-lipoxygenase inhibitors, cromolyn) must be stable for 30 days before screening, and continue without dosage changes throughout study.
* The patient has a blood eosinophil count of at least 400/μL.
* Female patients must be surgically sterile, 2 years postmenopausal, or must have a negative pregnancy test ßHCG at screening (serum) and baseline (urine).
* Female patients of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after the end-of-treatment visit. Acceptable methods of contraception include barrier method with spermicide, abstinence, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected).
* Written informed consent is obtained. Patients 12 through 17 years old, where participating, need to provide assent in accordance with local standards.
* Other inclusion criteria apply.

Exclusion Criteria:

* The patient has a clinically meaningful comorbidity that would interfere with the study schedule or procedures, or compromise the patient's safety.
* The patient has known hypereosinophilic syndrome (HES).
* The patient has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease, pulmonary fibrosis, or lung cancer). The patient has other pulmonary conditions with symptoms of asthma and blood eosinophilia (eg, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis).
* The patient is a current smoker (ie, has smoked within the last 6 months prior to screening).
* The patient has a history of use of systemic immunosuppressive or immunomodulating agents (anti-IgE mAb, methotrexate, cyclosporin, interferon-α, or anti-tumor necrosis factor mAb) within 6 months prior to study entry (screening).
* The patient is currently using systemic corticosteroids (includes use of oral corticosteroids).
* The patient has a current infection or disease that may preclude assessment of asthma.
* The patient is expected to be poorly compliant with study drug administration, study procedures, or visits.
* The patient has any aggravating factors that are inadequately controlled (eg, gastroesophageal reflux disease).
* The patient has participated in any investigative drug or device study within 30 days prior to screening.
* The patient has participated in any investigative biologics study within 90 days prior to screening.
* The patient has previously received anti-hIL-5 monoclonal antibody (eg, mepolizumab).
* Female patients who are pregnant, or nursing, or, if of childbearing potential and not using a medically accepted, effective method of birth control (e.g. spermicide, abstinence, IUD, or steroidal contraceptive [oral, transdermal, implanted, and injected]) are excluded from this study.
* The patient has a current infection or disease that may preclude assessment of asthma.
* The patient has a history of concurrent immunodeficiency (human immunodeficiency, acquired immunodeficiency syndrome, or congenital immunodeficiency). Patients in Argentina must have documented serology testing for HIV performed during screening.
* Other exclusion criteria apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Senior Director - Worldwide Clinical Research, MD, Study Director — Cephalon
Locations (89):
- United States (26):
  - Teva Investigational Site 12, Anaheim, California
  - Teva Investigational Site 11, Fountain Valley, California
  - Teva Investigational Site 43, Los Angeles, California
  - Teva Investigational Site 4, Orange, California
  - Teva Investigational Site 15, Walnut Creek, California
  - Teva Investigational Site 2, Colorado Springs, Colorado
  - Teva Investigational Site 24, Largo, Florida
  - Teva Investigational Site 27, Miami, Florida
  - Teva Investigational Site 5, Miami, Florida
  - Teva Investigational Site 19, Tallahassee, Florida
  - Teva Investigational Site 17, Trinity, Florida
  - Teva Investigational Site 18, Valrico, Florida
  - Teva Investigational Site 6, Lilburn, Georgia
  - Teva Investigational Site 3, Savannah, Georgia
  - Teva Investigational Site 7, Iowa City, Iowa
  - Teva Investigational Site 8, Omaha, Nebraska
  - Teva Investigational Site 26, Summit, New Jersey
  - Teva Investigational Site 20, Cincinnati, Ohio
  - Teva Investigational Site 1, Medford, Oregon
  - Teva Investigational Site 73, Lincoln, Rhode Island
  - Teva Investigational Site 9, Providence, Rhode Island
  - Teva Investigational Site 21, Charleston, South Carolina
  - Teva Investigational Site 16, Fort Worth, Texas
  - Teva Investigational Site 10, Houston, Texas
  - Teva Investigational Site 14, San Antonio, Texas
  - Teva Investigational Site 45, San Antonio, Texas
- Argentina (9):
  - Teva Investigational Site 121, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 126, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 127, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 128, Quilmes-Buenos Aires
  - Teva Investigational Site 125, Rosario
  - Teva Investigational Site 123, Rosario-Santa Fe
  - Teva Investigational Site 120, San Miguel de Tucuman - Tucuma
  - Teva Investigational Site 122, San Miguel de Tucuman - Tucuma
  - Teva Investigational Site 124, San Miguel de Tucuman - Tucuma
- Belgium (4):
  - Teva Investigational Site 261, Brussels
  - Teva Investigational Site 264, Brussels
  - Teva Investigational Site 260, Ghent
  - Teva Investigational Site 263, Liège
- Brazil (9):
  - Teva Investigational Site 146, Belo Horizonte
  - Teva Investigational Site 150, Florianópolis
  - Teva Investigational Site 140, Porto Alegre
  - Teva Investigational Site 143, Porto Alegre
  - Teva Investigational Site 144, Porto Alegre
  - Teva Investigational Site 145, Porto Alegre
  - Teva Investigational Site 147, Porto Alegre - RS
  - Teva Investigational Site 142, Santo André
  - Teva Investigational Site 141, São Paulo
- Canada (4):
  - Teva Investigational Site 103, Calgary
  - Teva Investigational Site 101, Montreal
  - Teva Investigational Site 104, Newmarket
  - Teva Investigational Site 105, Windsor
- Colombia (6):
  - Teva Investigational Site 181, Bogotá
  - Teva Investigational Site 184, Bogotá
  - Teva Investigational Site 185, Bogotá
  - Teva Investigational Site 182, Cali
  - Teva Investigational Site 180, Floridablanca
  - Teva Investigational Site 183, Medellín
- France (5):
  - Teva Investigational Site 343, Grenoble
  - Teva Investigational Site 342, Marseille
  - Teva Investigational Site 341, Montpellier
  - Teva Investigational Site 340, Nantes
  - Teva Investigational Site 344, Pessac
- Hungary (7):
  - Teva Investigational Site 401, Balassagyarmat
  - Teva Investigational Site 406, Edelény
  - Teva Investigational Site 400, Miskolc
  - Teva Investigational Site 404, Mosonmagyaróvár
  - Teva Investigational Site 403, Sopron
  - Teva Investigational Site 407, Százhalombatta
  - Teva Investigational Site 402, Tatabánya
- Israel (3):
  - Teva Investigational Site 422, Petah Tikva
  - Teva Investigational Site 421, Rehovot
  - Teva Investigational Site 420, Tel Aviv
- Mexico (5):
  - Teva Investigational Site 203, Distrito Federal
  - Teva Investigational Site 205, Distrito Federal
  - Teva Investigational Site 204, Guadalajara, JAL
  - Teva Investigational Site 200, Hermosillo, Sonora
  - Teva Investigational Site 202, Tijuana, B.C.
- Teva Investigational Site 460, Heerlen, Netherlands
- Poland (7):
  - Teva Investigational Site 507, Bialystok
  - Teva Investigational Site 513, Gdansk
  - Teva Investigational Site 512, Lodz
  - Teva Investigational Site 505, Lublin
  - Teva Investigational Site 500, Ostrów Wielkopolski
  - Teva Investigational Site 502, Sopot
  - Teva Investigational Site 504, Tarnów
- Sweden (3):
  - Teva Investigational Site 602, Gothenburg
  - Teva Investigational Site 600, Lund
  - Teva Investigational Site 601, Malmo

REFERENCES:
- [Derived] Bjermer L, Lemiere C, Maspero J, Weiss S, Zangrilli J, Germinaro M. Reslizumab for Inadequately Controlled Asthma With Elevated Blood Eosinophil Levels: A Randomized Phase 3 Study. Chest. 2016 Oct;150(4):789-798. doi: 10.1016/j.chest.2016.03.032. Epub 2016 Apr 4. PMID 27056586

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1025 patients screened at 80 centers in 12 countries (Argentina, Belgium, Brazil, Canada, Colombia, Hungary, Israel, Mexico, Netherlands, Poland, Sweden, and the US), 315 patients met entry criteria at 68 centers and were considered to be eligible for enrollment.
Period: Overall Study
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Started | 105 | 104 | 106
Safety Analysis Set | 105 | 103 | 103
Full Analysis Set | 105 | 103 | 103
Pharmacokinetic Analysis Set | 105 | 103 | 103
Completed | 85 | 92 | 88
Not Completed | 20 | 12 | 18
Not completed — Protocol Violation | 4 | 3 | 2
Not completed — Lack of Efficacy | 2 | 3 | 1
Not completed — Adverse Event | 9 | 1 | 7
Not completed — Withdrawal by Subject | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Other | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg | Total
Number analyzed (Participants) | 105 | 104 | 106 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (14.89) | 44.5 (14.03) | 43.0 (14.41) | 43.9 (14.42)
Age, Customized [Number; unit: participants]
  Adolescents (12-17 years) | 5 | 5 | 5 | 15
  Adults (18-64 years) | 93 | 91 | 99 | 283
  From 65-84 years | 7 | 8 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 62 | 183
  Male | 43 | 45 | 44 | 132
Race/Ethnicity, Customized [Number; unit: participants]
  White | 85 | 80 | 90 | 255
  Black | 7 | 6 | 5 | 18
  Asian | 0 | 2 | 2 | 4
  American Indian or Alaskan Native | 1 | 0 | 0 | 1
  Pacific Islander | 1 | 0 | 0 | 1
  Other | 11 | 16 | 9 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 29 | 29 | 31 | 89
  Non-Hispanic and Non-Latino | 74 | 73 | 75 | 222
  Unknown | 2 | 2 | 0 | 4
Asthma Exacerbation Within the Last 12 Months [Number; unit: participants] — A stratification factor with data as reported in the case report form
  participants
    Yes | 57 | 58 | 60 | 175
    No | 48 | 46 | 46 | 140
Weight [Mean (Standard Deviation); unit: kg] | 77.0 (20.1) | 75.9 (18.8) | 75.7 (20.3) | 76.2 (19.70)
Height [Mean (Standard Deviation); unit: cm] | 166.4 (10.93) | 166.2 (12.21) | 165.9 (10.24) | 166.2 (11.12)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (6.01) | 27.6 (6.68) | 27.4 (6.87) | 27.6 (6.51)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Forced Expiratory Volume In 1 Second (FEV1) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer. The during treatment (weeks 4, 8, 12 and 16) average FEV1 was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Day 0 (baseline, pre-dose), Weeks 4, 8, 12 and 16
Population: Full analysis set-all patients randomly assigned to treatment and treated with at least 1 dose of study drug. Number of participants analyzed includes those who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 102
liters | 0.126 (0.0549) | 0.242 (0.0556) | 0.286 (0.0548)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; The primary variable was analyzed using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — The overall treatment effect for each reslizumab dose was compared to placebo using a 2-sided t-test at the a priori significance level of 0.05; Mean Difference (Final Values) = 0.160, 95% CI 2-sided [0.060 to 0.259], Standard Error of Mean 0.0507
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0237, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI 2-sided [0.016 to 0.215], Standard Error of Mean 0.0508

2. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The FVC is the volume of air that can be forcibly blown out after full inspiration, measured in liters. The during treatment (weeks 4, 8, 12 and 16) average FVC was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set. Number of participants analyzed includes those who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 102
liters | 0.172 (0.0614) | 0.220 (0.0623) | 0.301 (0.0613)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; As with the primary outcome, this respiratory test outcome was analyzed using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements; Test type: Superiority or Other; p = 0.0174, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [0.023 to 0.237], Standard Error of Mean 0.0543
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3731, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.058 to 0.155], Standard Error of Mean 0.0543

3. Secondary Outcome: Change From Baseline in Forced Expiratory Flow at 25% to 75% Forced Vital Capacity (FEF 25%-75%) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The FEF 25%-75% is the force expiratory flow at 25% to 75% of the Forced Vital Capacity (FVC). The during treatment (weeks 4, 8, 12 and 16) average FEF 25%-75% was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set. Number of participants analyzed includes those who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 102
liters/second | -0.145 (0.1342) | -0.114 (0.1361) | 0.089 (0.1342)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0552, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.233, 95% CI 2-sided [-0.005 to 0.472], Standard Error of Mean 0.1212
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.209 to 0.270], Standard Error of Mean 0.1215

4. Secondary Outcome: Change From Baseline in % Predicted Expiratory Volume In 1 Second (FEV1) at Week 16 and at Endpoint
Description: The percent predicted FEV1 is the ratio of the volume of air expired in the first second of a forced expiration to the patient's predicted FEV based on a similar population without asthma. Endpoint =week 16 or early withdrawal.
Time Frame: Day 1 (baseline, pre-dose), Week 16, endpoint
Population: Full analysis set of participants with assessments at stated timeframes.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 102
percentage of predicted FEV1
  Week 16 (n=84, 92, 91) | 0.8 (11.92) | 4.9 (15.06) | 7.5 (14.74)
  Endpoint (n=103, 101, 102) | 0.8 (13.83) | 5.5 (15.16) | 6.7 (15.01)

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A higher score is an indication of poorer asthma control. The during treatment (weeks 4, 8, 12 and 16) average ACQ was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 101
units on a scale | -0.494 (0.1231) | -0.732 (0.1250) | -0.853 (0.1233)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.359, 95% CI 2-sided [-0.577 to -0.140], Standard Error of Mean 0.1110
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0329, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.238, 95% CI 2-sided [-0.456 to -0.019], Standard Error of Mean 0.1108

6. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) at Week 16 or at Last Observed Value
Description: The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses. Five of the activity questions were "patient-specific," which means that each patient identified and scored 5 activities in which the patient was limited by asthma; these 5 activities were identified at the first visit and retained for all subsequent follow-up visits.
  Positive change from baseline scores indicate improvement in quality of life. The AQLQ score was only assessed once during the study at week 16 or at early withdrawal, i.e. last postbaseline assessment if within 3 to 5 weeks of the last dose of study drug.
Time Frame: Day 1 (baseline, pre-dose), Week 16 or last observed value
Population: Full analysis set of participants with assessments at stated timeframes.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 101 | 96 | 99
units on a scale | 0.779 (0.1817) | 1.057 (0.1881) | 1.138 (0.1829)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0241, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.359, 95% CI 2-sided [0.047 to 0.670], Standard Error of Mean 0.1582
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0822, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.278, 95% CI 2-sided [-0.036 to 0.591], Standard Error of Mean 0.1591

7. Secondary Outcome: Change From Baseline in Asthma Symptom Utility Index (ASUI) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control. The during treatment (weeks 4, 8, 12 and 16) average ASUI was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Positive change from baseline values indicate improvement in asthma symptoms. Information was obtained from questionnaire about asthma symptoms.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set, including patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 101
units on a scale | 0.082 (0.0218) | 0.132 (0.0221) | 0.129 (0.0218)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0160, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [0.009 to 0.085], Standard Error of Mean 0.0193
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.051, 95% CI 2-sided [0.012 to 0.089], Standard Error of Mean 0.0193

8. Secondary Outcome: Change From Baseline in Short-Acting Beta-Agonist (SABA) Use Over 16 Weeks Using Mixed Model for Repeated Measures
Description: SABA are used for quick relief of asthma symptoms. To measure SABA use, at each clinical visit patients were asked to recall their usage of SABA therapy within the last 3 days of the scheduled visit. If usage was confirmed, the number of puffs used was recorded. For the purpose of summaries, an average daily usage was evaluated by dividing the total number of puffs recorded over 3 days by 3.
  The during treatment (weeks 4, 8, 12 and 16) average SABA use was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set, including patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: SABA puffs per day
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 102 | 101 | 102
SABA puffs per day | -0.3 (0.28) | -1.0 (0.28) | -0.9 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0151, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.624, 95% CI 2-sided [-1.126 to -0.121], Standard Error of Mean 0.2551
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0119, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.648, 95% CI 2-sided [-1.152 to -0.144], Standard Error of Mean 0.2559

9. Secondary Outcome: Change From Baseline in Blood Eosinophil Count Over 16 Weeks Using Mixed Model for Repeated Measures
Description: Blood eosinophil counts were measured using a standard complete blood count (CBC) with differential blood test at each scheduled visit, and from all patients experiencing a serious adverse event, an adverse event leading to withdrawal, or an exacerbation of asthma symptoms. The during treatment (weeks 4, 8, 12 and 16) average eosinophil counts were estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline values correlate to reduced asthma severity.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Full analysis set, including patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: 10^9 blood eosinophil/L
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 103 | 101 | 102
10^9 blood eosinophil/L | -0.035 (0.0271) | -0.358 (0.0277) | -0.529 (0.0270)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab - 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0000, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.494, 95% CI 2-sided [-0.542 to -0.447], Standard Error of Mean 0.0242
Statistical Analysis 2: Comparison: Placebo vs Reslizumab - 0.3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0000, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.323, 95% CI 2-sided [-0.370 to -0.275], Standard Error of Mean 0.0243

10. Secondary Outcome: Participants With Adverse Events
Description: An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes. The last postbaseline value for approximately 10 patients in each treatment group is the 90-day follow-up visit post end-of-treatment (approx. Week 29).
Time Frame: Day 1 (post-dose) to Week 29
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 105 | 103 | 103
participants
  At least 1 AE | 66 | 59 | 61
  Severe AE | 4 | 2 | 7
  Treatment-related AE | 8 | 6 | 12
  Withdrawn from study due to AE | 10 | 1 | 6
  Withdrawn due to treatment-related AE | 0 | 0 | 1
  Death | 0 | 0 | 0
  Serious AE (excluding death outcome) | 1 | 0 | 4
  Treatment-related serious AEs | 0 | 0 | 0

11. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Abnormal Lab Values
Description: Data represents participants with potentially clinically significant (PCS) abnormal serum chemistry, hematology (except for eosinophil values), and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * GGT = gamma-glutamyl transpeptidase: >= 3*upper limit of normal. Normal range is 5-49 U/L.
  * Total bilirubin: >=34.2 μmol/L
  * White blood cells: <=3.0 10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 %
  * Platelets: >=700 10^9/L
  * Absolute neutrophil count: <=1.0 10^9/L
  * Urinalysis: blood, glucose, ketones and total protein: >=2 unit increase from baseline
  The last postbaseline value for approximately 10 patients in each treatment group is the 90-day follow-up visit post end-of-treatment (approx. Week 29).
Time Frame: Day 2 to Week 29
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 105 | 103 | 103
participants
  >=1 PCS abnormal serum chemistry value | 1 | 5 | 2
  Blood urea nitrogen | 0 | 0 | 1
  Creatinine | 1 | 0 | 0
  Uric acid | 0 | 0 | 2
  GGT | 0 | 4 | 0
  Total bilirubin | 0 | 1 | 0
  >=1 PCS abnormal hematology value | 4 | 7 | 3
  White blood cells | 0 | 0 | 1
  Hemoglobin | 0 | 2 | 0
  Hematocrit | 2 | 6 | 2
  Platelets | 0 | 0 | 1
  Absolute neutrophil count | 2 | 1 | 0
  >=1 PCS abnormal urinalysis value | 21 | 21 | 18
  Blood in urine | 10 | 11 | 6
  Glucose in urine | 3 | 4 | 5
  Ketones in urine | 0 | 1 | 3
  Total protein in urine | 11 | 11 | 11

12. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Vital Signs Values
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Sitting pulse - high: >100 and increase of >= 30 beats/minute
  * Sitting pulse - low: <50 and decrease of >=30 beats/minute
  * Sitting diastolic blood pressure: >100 and increase of >=12 mmHg
  * Respiration rate: >24 and increase of >=10 breaths/minute
  * Body temperature: <96.5° Fahrenheit or <35.8° Celsius
  The last postbaseline value for approximately 10 patients in each treatment group is the 90-day follow-up visit post end-of-treatment (approx. Week 29).
Time Frame: Day 2 to Week 29
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 105 | 103 | 103
participants
  >=1 PCS abnormal vital sign | 12 | 16 | 16
  Sitting pulse - high | 0 | 1 | 2
  Sitting pulse - low | 0 | 1 | 1
  Sitting diastolic blood pressure - high | 0 | 0 | 1
  Respiration rate - high | 0 | 2 | 0
  Body temperature - low | 12 | 13 | 13

13. Secondary Outcome: Shifts From Baseline to Endpoint in Electrocardiogram Findings
Description: Participant counts in each category of shift from baseline to endpoint of ECG finding. Findings summarized as normal or abnormal.
Time Frame: Weeks -4 to -2 (Screening Visit), Week 16
Population: Safety analysis set of participants with both baseline and endpoint values.
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 102 | 99 | 101
participants
  Normal to Normal | 64 | 70 | 63
  Normal to Abnormal | 14 | 10 | 15
  Abnormal to Normal | 11 | 9 | 13
  Abnormal to Abnormal | 13 | 10 | 10

14. Secondary Outcome: Participants With a Positive Anti-Reslizumab Antibody Status at Baseline, Week 8, Week 16, Endpoint, and Overall
Description: Counts of participants with a positive anti-drug antibody (ADA) response during treatment is offered for the two experimental treatment arms. Blood samples were collected for determination of ADAs before study drug infusion at baseline, visit 4 (week 8), and at visit 6 (week 16: EOT or early withdrawal) from patients in all 3 treatment groups (ie, placebo, 0.3 mg/kg reslizumab, and 3.0 mg/kg reslizumab); however, only the blood samples drawn from patients treated with either 0.3 mg/kg reslizumab or 3.0 mg/kg reslizumab were analyzed. Serum samples from patients who were treated with reslizumab were analyzed for ADA by Teva (Teva Biopharmaceuticals USA, Rockville, MD) using a validated homogeneous solution-based bridging enzyme-linked immunosorbent assay (ELISA).
  Endpoint =week 16 or early withdrawal.
Time Frame: Day 1 (pre-dose), week 8, 16 and endpoint
Population: Pharmacokinetic analysis set. Anti-Reslizumab antibody status was not analyzed for patients in the Placebo treatment arm.
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Number analyzed (Participants) | 0 | 103 | 103
participants
  Overall (n=102, 103) |  | 12 | 11
  Baseline (n=99, 98) |  | 8 | 8
  Week 8 (n=90, 94) |  | 8 | 10
  Week 16 (n=91, 89) |  | 7 | 5
  Endpoint (n=101, 102) |  | 10 | 6

ADVERSE EVENTS:
Time Frame: Day 1 to Week 29. The last postbaseline value for approximately 10 patients in each treatment group is the 90-day follow-up visit post end-of-treatment (approx. Week 29). Events reported during the followup were treated as treatment-emergent.
Arm/Group | Placebo | Reslizumab - 0.3 mg/kg | Reslizumab - 3.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/103 | 4/103
Other Adverse Events (participants affected / at risk) | 28/105 | 20/103 | 28/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | Reslizumab - 0.3 mg/kg (N=103) | Reslizumab - 3.0 mg/kg (N=103)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | Reslizumab - 0.3 mg/kg (N=103) | Reslizumab - 3.0 mg/kg (N=103)
Nasopharyngitis (Infections and infestations) | 4 (5) | 6 (9) | 6 (6)
Headache (Nervous system disorders) | 6 (7) | 8 (9) | 11 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 6 (10) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.